CLINICAL TRIAL: NCT00854022
Title: Genetic Susceptibility to Renal Cell Carcinoma
Brief Title: Genetic Susceptibility to Kidney Cancer
Status: Terminated | Type: Observational
Why Stopped: Funding ended
Sponsor: Baylor College of Medicine (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Seth Lerner, Professor, Baylor College of Medicine
Other Study IDs: H-17150
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will utilize the blood collected to run several laboratory analyses that will assess DNA damage/repair, telomere length, telomerase activity, and other genetic instability as predictors of RCC risk. All information linking this unique identifier to the participant will be kept in a secure location under lock-and-key password protected.
  In addition, RCC tumor and adjacent normal tissue samples may be obtained from the MDACC Institutional Tissue Bank (ITB) for cases only. The samples obtained will be left over from surgical procedures, so as to prevent any additional distress to the patient.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy: Healthy adults, of any ethnicity, or sex, and with no previous history of cancer, except for non-melanoma skin cancer
- RCC: Adult patients with newly diagnosed (diagnosed within the year of enrollment) renal carcinoma (RCC) any ethnicity, or sex, who have not received prior chemotherapy or radiotherapy.

SUMMARY:
This study will further the understanding of the genetic events leading to the development of RCC.

DETAILED DESCRIPTION:
This study will further the understanding of the genetic events leading to the development of RCC; explore the genetic basis for genetic instability and how it affects cancer risk; and eventually provide a means of identifying a subgroup of individuals who are most likely to develop RCC. Such individuals may then be targeted for intervention programs such as chemoprevention or dietary modification.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of any ethnicity or sex, who have a been diagnosed with possible Renal Cell Carcinoma within the past year.

Exclusion Criteria:

* Must not have received chemotherapy, biological therapy or radiation therapy in the 6 months preceding enrollment will
* Must not have had RCC, or metastatic RCC,
* Must not have had a renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with newly diagnosed (diagnosed within the year of enrollment) with possible Renal Cell Carcinoma (RCC)
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To identify interindividual differences in inherited genetic instability | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Seth P. Lerner, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States